CLINICAL TRIAL: NCT02865954
Title: Use of Iball Mobile Health Technology in Pelvic Floor Muscle Training in the Postpartum Period: a Pilot Mixed Methods Study
Brief Title: Iball & Pelvic Floor Muscle Training
Acronym: iball
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sinead Dufour, Assistant Clinical Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: iball_McMaster
Record Dates: First submitted 2016-07-27; First posted 2016-08-15 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Segmental Dysfunction of the Pelvic Region

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iball intervention (Experimental): Use of iball pelvic floor training mhealth application for 16 weeks.
  Interventions: Device: iball (mhealth application)
- Standard Care (No Intervention): Standard Care - control group

INTERVENTIONS:
Device: iball (mhealth application) — mhealth application and associated device to support activation of the pelvic floor muscles.
  Arms: iball intervention

SUMMARY:
he postpartum period is vulnerable to dysfunction of the pelvic floor musculature, which is associated with incontinence, pain, reduced stability of the core and functional deficits. The Society of Obstetricians and Gynaecologists of Canada recommends instruction on the correct performance of pelvic floor muscle exercises, commonly known as Kegels, as standard care. However, only a small proportion of women seek medical care for incontinence in Canada. Recently, there has been an influx of mobile Health technology applications marketed for pelvic floor restoration and fitness that have not been studied. The existence of mHealth technologies may represent an innovative mode to support pelvic health, however systematic exploration to substantiate claims and proposed benefit is required. This pilot study aims to understand the utility of a new mobile health application, iball, as a rehabilitation tool to promote optimal pelvic floor function and to correct pregnancy related pelvic floor dysfunction. The iball is comprised of a device and a mobile app, and it has been brought to market in Europe as a consumer product. The study aims to assess the acceptability, feasibility, and effectiveness of the iball as a pelvic floor muscle training intervention, in comparison to standard care.

DETAILED DESCRIPTION:
Participants would be recruited through three midwifery practices: 1) The Hamilton Midwives; 2) Burlington & Area Midwives Inc.; and 3) Community Midwives of Halton. Women in the third trimester of their first pregnancy, presenting at these sites will be invited to participate. The goal is to enrol a heterogeneous sample of pregnant women in the Hamilton-Halton region.

A two-step strategy will be used to recruit study participants. First, recruiting sites will attend an information session related to the study. Recruitment posters with tear-off tabs containing the study email (iballstudy@gmail.com) will be posted at the sites. Interested participants will contact the study co-ordinator. Over the phone, the study co-ordinator will determine that the patient is eligible, review the letter of information with the patient, and schedule them for a baseline assessment at approximately 6-weeks post-partum. The letter of information will be emailed to the patient so that they may follow along during the review. All Internet transmission will be performed on campus through MacSecure, or performed off campus through a Virtual Private Network (VPN) provided by McMaster University.

The patient will provide informed, written consent at the baseline appointment and prior to the assessment.

The study compares a 16-week iball pelvic floor training protocol to a 16-week standard care regimen. Sixty participants will be recruited and randomly assigned to the standard care (control) group or the iball intervention group. All participants will meet with an assessor (Dr. Sinead Dufour or Dr. Donna Fedorkow) to undergo a pre-and a post-intervention assessment. Each assessment (30min) will consist of a (15min) internal pelvic exam, following the PERFECT criteria, and two (15min) self-report questionnaires, the Urogenital Distress Inventory-Short Form (UDI-6) and the Incontinence Impact Questionnaire-Short Form (IIQ-7). The pre-study assessment will take place approximately 6 weeks post-partum. The post-study assessment will take place at the end of the 16-week study period. At 8 weeks, midway through the intervention period, all participants will be emailed by the study co-ordinator as a means to provide any support that might be needed.

At the pre-study assessment, the standard care group will receive instructions on how to perform a correct pelvic floor contraction through a digital pelvic examination. In addition to receiving the same standard care instructions, the iball intervention group will undergo a training session (15min) on how to use the iball device and app with the research co-ordinator.

The post-study assessment will require additional time from both groups. The standard care group will answer three self-administered close-ended questions (5min). In addition to answering two of the three close-ended questions (5min), the intervention group will also participate in a semi-structured interview (30min) with the research assistant either in-person or over the phone, depending on the participant's preference.

ELIGIBILITY:
Inclusion Criteria:

* Women in their third trimester, first pregnancy.

Exclusion Criteria:

* Currently seeing a pelvic health physiotherapists or participating in a pelvic floor fitness program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the iball intervention (via qualitative data collection) | 16 weeks
  1. Tell me about your experiences using the iball device?
  2. What aspects of iball were the most useful or helpful?
  3. Which aspects of iball were least useful or helpful?
  4. Are there any changes you would make to the iball device or app?
  5. If you had to explain iball to friend, what would you say?
  6. Would you recommend it to a friend - why or why not?
  7. Do you plan on continuing to use iball at this time? Why or why not?
  8. Would you consider using iball again in the future?

SECONDARY OUTCOMES:
PERFECT - pelvic floor exam scores | 16 weeks
Urinary Distress Inventory (UDI-6) | 16 weeks
  Standardized outcome measure
Incontinence Impact Questionnaire (IIQ-7) | 16 weeks
  Standardized outcome measure

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735
- [Derived] Dufour S, Fedorkow D, Kun J, Deng SX, Fang Q. Exploring the Impact of a Mobile Health Solution for Postpartum Pelvic Floor Muscle Training: Pilot Randomized Controlled Feasibility Study. JMIR Mhealth Uhealth. 2019 Jul 11;7(7):e12587. doi: 10.2196/12587. PMID 31298221